CLINICAL TRIAL: NCT00818168
Title: Remicade Safety Line (Ankylosing Spondylitis)
Brief Title: Remicade Safety Line (Ankylosing Spondylitis)(Study P03275)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P03275
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab: Subjects with ankylosing spondylitis who were treated with infliximab. The dosage and infusion intervals were employed in accordance to the Summary of Product Characteristics (SmPC)
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Dosage and infusion intervals were employed in
  accordance to the Summary of Product Characteristics (SmPC)
  Other Names: Remicade; SCH 215596

SUMMARY:
This observational study is in line with the German educational plan with the aim to implement a tool to increase and monitor the awareness of tuberculosis screening and to reinforce the patient eligibility for a treatment with Remicade according to the Summary of Product Characteristics (SmPc).

DETAILED DESCRIPTION:
This study population was chosen from a non-probability sample.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with ankylosing spondylitis.

Exclusion Criteria:

* As per Summary of Product Characteristics (SmPC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with ankylosing spondylitis.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2003-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were those with Ankylosing spondylitis (AS) starting treatment with Remicade at 26 sites in Germany from Jul 2003 through Dec 2010
Period: Overall Study
Arm/Group | Infliximab
Started | 320
Completed | 250 (Includes 78 participants whose completer/non-completer status was not reported (missing))
Not Completed | 70
Not completed — Lack of Efficacy | 18
Not completed — Pregnancy | 2
Not completed — Withdrawal by Subject | 16
Not completed — Lost to Follow-up | 7
Not completed — Adverse Event | 19
Not completed — Reason for Non-completion Not reported | 6
Not completed — Participant Moved | 2

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.99 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 210
Region of Enrollment [Number; unit: participants]
  Germany | 320

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had the Mendel Mantoux Test as the First Screening Test for Active or Latent Tuberculosis (TB) Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the Mendel Mantoux test (tuberculin sensitivity skin test by intradermal injection) as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing (represents no entry, but may mean another test was performed as first screening test and documented)
Time Frame: Baseline
Population: Data was analyzed for all AS patients whose data was entered into the database and finalized by signature of the physician.
Measure: Number; unit: participants
Arm/Group | Infliximab
Number analyzed (Participants) | 320
participants
  Yes | 310
  No | 9
  Missing | 1

2. Primary Outcome: Number of Participants Who Had the Tine Test as the First Screening Test for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the Tine test (multiple puncture tuberculin skin test) as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing (represents no entry, but may mean another test was performed as first screening test and documented)
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 320
Participants
  Yes | 8
  No | 311
  Missing | 1

3. Primary Outcome: Number of Participants Who Had the In-vitro TB Test as the First Screening Test for Active or Latent Tuberculosis Before Starting
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the in-vitro TB test (cellular blood test, i.e. gamma interferon release assays) as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing (represents no entry, but may mean another test was performed as first screening test and documented)
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 320
Participants
  Yes | 9
  No | 154
  Missing | 157

4. Primary Outcome: Number of Participants Who Had a Chest X-ray as Part of TB Screening for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). If done according to guidelines, complete TB screening comprised a TB screening test and a chest X-ray. The number of participants who had a frontal chest X-ray was presented in three categories:
  * Yes
  * No
  * Missing
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 320
Participants
  Yes | 290
  No | 29
  Missing | 1

5. Secondary Outcome: Assessment of Disease Activity by Means of the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at the Time of Enrollment and at the First Infusion
Description: The BASDAI score was calculated based on the responses to questions 1-6, with each component rated on a scale of 0 (best) to 10 (worst) based on the severity of various characteristics. A decrease in BASDAI over time indicated improvement in disease activity. The score corresponded to the sum of the point values from questions 1-4 and the mean of the point values from questions 5 and 6, subsequently divided by five. BASDAI was calculated at the time of enrollment (baseline) and at the time of first infusion.
Time Frame: Baseline and time of first infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 320
Units on a scale
  BASDAI at Time of Enrollment (n=268) | 5.15 (2.14)
  BASDAI at First Infusion (n=82) | 5.19 (2.35)

ADVERSE EVENTS:
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 2/320
Other Adverse Events (participants affected / at risk) | 0/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=320)
anaphylactic shock (Immune system disorders) | 1 (1)
lupus-like disease (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results belong to the SPONSOR only, all investigators are not allowed to publish trial results without permission of the SPONSOR.